CLINICAL TRIAL: NCT04457999
Title: Clinical Outcome of Lipiflow Treatment Prior to Cataract Surgery in Dry Eye Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, M.D. Ph.D, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-03-011
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipiflow treatment (Experimental): Lipiflow thermal pulsation prior to cataract surgery
  Interventions: Device: Lipiflow Thermal pulsation

INTERVENTIONS:
Device: Lipiflow Thermal pulsation — Single vectored thermal pulsation treatment for dry eye

SUMMARY:
To investigate the clinical outcome of Lipiflow treatment prior to cataract surgery in patients with meibomian gland dysfunction and dry eye disease

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 21, who will get catarct surgeyr
* Patients whose visual acuity anticipated better than 20/25 after surgery
* Patients with informed consent
* Patients with meibomian gland dysfunction

Exclusion Criteria:

* ocular injury, active injection
* uncontrolled systemic disease
* Contact lens wear within 1 month
* Allergic to fluorescein sodium or topical anesthetics
* ocular surgery or trauma within 6 months
* disorder of lid anatomy
* other reason for decreased vision other than cataract
* anticipated visual acuity less than 20/25
* Patients less than 20 years.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-07-02 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
improvement of dry eye symptom | 1 month
  ocular dryness

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No